CLINICAL TRIAL: NCT00344058
Title: Abbreviated Post-partum Magnesium Sulfate Seizure Prophylaxis in Preeclampsia: A Comparison of 12 and 24 Hour Regimens
Brief Title: Abbreviated MgSO4 Therapy in Post-partum Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 01001-OBG-01
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy; Preeclampsia
Keywords: pregnancy; preeclampsia; treatment
MeSH Terms: conditions — Pre-Eclampsia

INTERVENTIONS:
Drug: abbreviation of magnesium sulfate therapy (12 hours versus the traditional 24 hours after delivery)

SUMMARY:
Magnesium sulfate is used for seizure prophylaxis in pregnancies complicated by preeclampsia. There is debate as to how long to continue this therapy after delivery of the pregnancy. Different schemes have been offered to shorten the exposure to magnesium sulfate after delivery, with little data. We seek to investigate the effect of shortened magnesium sulfate therapy on the post-partum recovery phase of mild preeclampsia. Our hypothesis was that shortened therapy (12 hours versus the traditional 24 hours post-partum) has no effect on disease course, and will result in significantly shorter exposure to magnesium sulfate.

DETAILED DESCRIPTION:
The study has been completed at this time.

Consenting women with suspected mild preeclampsia (new onset/exacerbated hypertension with proteinuria) were randomly assigned 12 (12-hour) or 24-hours (24-hour) of postpartum MgSO4. Treatment was continued beyond the initially assigned time period for new findings of severe preeclampsia. Clinical and laboratory data were collected. Analysis was by intent to treat, utilizing Fisher's exact, chi-square, and Student's t-tests where appropriate

ELIGIBILITY:
Inclusion Criteria:

* Women with suspected mild preeclampsia diagnosed antepartum, intrapartum, or post-partum were eligible for inclusion after delivery at term (≥ 34 weeks' gestational age).

Exclusion Criteria:

* Inability to give informed consent, preterm delivery, severe preeclampsia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2001-01 (Actual); Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Time of magnesium sulfate therapy (minutes)
Blood pressure
Maternal symptoms (headaches, blurred vision, chest pain, shortness of breath)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh M Ehrenberg, MD, Principal Investigator — MetroHealth Medical Center at Case Western Reserve School of Medicine
Locations (1):
- MetroHealth Medical Center, Labor and Delivery, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Ehrenberg HM, Mercer BM. Abbreviated postpartum magnesium sulfate therapy for women with mild preeclampsia: a randomized controlled trial. Obstet Gynecol. 2006 Oct;108(4):833-8. doi: 10.1097/01.AOG.0000236493.35347.d8. PMID 17012443